CLINICAL TRIAL: NCT03448510
Title: The Safety and Efficacy of Irreversible Electroporation Versus Standard Medication for the Treatment of Benign Prostatic Obstruction: a Randomized Controlled Trial
Brief Title: Irreversible Electroporation Versus Standard Medication for Benign Prostatic Obstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Yinghao Sun, MD, PhD, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRE-2018
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: lower urinary tract symptoms; male; benign prostatic obstruction; irreversible electroporation; urodynamics
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: Irreversible electroporation (IRE) is a novel ablation modality using electric pulses to create nanoscale defects in the cell membrane.
Who Masked: Outcomes Assessor
Masking Description: The data will be analyzed in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irreversible electroporation treatment (Experimental): Subjects will receive irreversible electroporation of the prostate
  Interventions: Device: Irreversible electroporation
- standard medication group (Active Comparator): Subjects will receive either α-blocker or 5α reductase monotherapy or combination therapy.
  Interventions: Drug: Standard Medication

INTERVENTIONS:
Device: Irreversible electroporation — The subject will receive Irreversible electroporation procedure which is a novel ablation modality using electric pulses to create nanoscale defects in the cell membrane.
  Arms: Irreversible electroporation treatment
Drug: Standard Medication — The subject will be prescribed with α-blocker or/and 5α-reductase inhibitors.
  Arms: standard medication group

SUMMARY:
Irreversible electroporation (IRE) is a novel ablation modality using electric pulses to create nanoscale defects in the cell membrane. It has been verified to be safe on the treatment of prostate, lung, liver and kidney masses. The present is a randomized, controlled trial, with a main purpose of looking into the safety and feasibility of irreversible electroporation for patients with benign prostatic obstruction.

DETAILED DESCRIPTION:
Benign prostatic obstruction (BPO) is the main reason to cause lower urinary tract symptoms (LUTS) in aged male. Oral medications, such as,α1-adrenoceptor antagonist and 5α-reductase inhibitors are the mainstay treatment options. However, some patients can not tolerate long-term use, due to either side effects or limited efficacy. Though transurethral resection or enucleation of prostate usually achieve significant symptom improvement, it's an end stage procedure and it is only reserved for carefully selected patients.

The development of focal ablative therapy yields minimally invasive treatment option for primary tumors such as the liver, lung, pancreas, kidney, and prostate. Among the novel techniques are cryoablation, radiofrequency ablation (RFA), microwave ablation, and high-intensity focused ultrasonography. Irreversible electroporation (IRE) is a one of the ablation modalities using electric pulses to create nanoscale defects in the cell membrane. IRE is not dependent on thermal energy and is therefore causing minimum damage to the blood vessels, nerves and tissue architecture. The present is a randomized, controlled trial, with a main purpose of looking into the safety and feasibility of irreversible electroporation for patients with benign prostatic obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 45 years or older.
2. The presence of voiding symptoms, i.e. slow stream, intermittent stream, hesitancy, straining, etc.
3. Qmax ≥ 5 mL/s and ≤ 15 mL/s with minimum voided volume of 125 mL or more during flow study.
4. The presence of bladder outlet obstruction during pressure-flow study.
5. International Prostatic Symptom Score (IPSS) ≥ 12 at screening.
6. Prostate volume ≥ 30 ml (using a transrectal ultrasound approach).
7. Total serum prostatic specific antigen (PSA) ≥ 1.5 ng/mL and ≤ 10 ng/mL at screening.
8. Subject is able to communicate and complete the questionnaires properly.
9. Written informed consent.

Exclusion Criteria:

1. Diagnosis or suspicion of bladder, prostate, urethral or pelvic tumor.
2. Patients with arrhythmia or history of cardiac pacemaker implantation.
3. Known lower urinary tract or pelvic surgical history.
4. Voiding symptoms as a result of urethral stricture, stone diseases, chronic prostatitis, space-occupying lesions etc.
5. Known neurogenic or congenital lower urinary tract dysfunction.
6. Rigid or flexible cystoscopy examination within the past 7 days at screening.
7. Existence of anatomical abnormalities of the urinary tract (e.g. diverticulum of the bladder or urethra, ectopic ureteral orifice etc.).
8. The presence of acute conditions, such as, urinary tract infection, fever, heart failure etc.
9. Patients with poor compliance or cognitive competence.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
The changes of maximum flow rate (ml/s) between baseline and during follow-up | Measured at baseline and 1, 3, 6 months during follow-up
  Maximum flow rate will be measured using urinary flow study

SECONDARY OUTCOMES:
The changes of IPSS scores between baseline and during follow-up | Measured at baseline and 1, 3, 6 months during follow-up
  Measured using a standard IPSS scoring system
The changes of IIEF scores between baseline and during follow-up | Measured at baseline and 1, 3, 6 months during follow-up
  Measured using a standard IIEF scoring system
The changes of maximum detrusor pressure at maximum flow rate between baseline and during follow-up | Measured at baseline and 3, 6 months during follow-up
  The data will be captured during pressure flow study
The changes of post void residual volume (ml) between baseline and follow-up | Measured at baseline and 1, 3, 6 months during follow-up
  Post void residual volume (ml) will be measured via ultrasound
The changes of prostate volume (ml) between baseline and follow-up | Measured at baseline and 1, 3, 6 during follow-up
  Prostate volume (ml) will be measured using transrectal prostate ultrasound and calculated as: prostate volume (ml) = length (mm) * width (mm) * height (mm) * 0.52.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagstaff PG, Buijs M, van den Bos W, de Bruin DM, Zondervan PJ, de la Rosette JJ, Laguna Pes MP. Irreversible electroporation: state of the art. Onco Targets Ther. 2016 Apr 22;9:2437-46. doi: 10.2147/OTT.S88086. eCollection 2016. PMID 27217767

DOCUMENTS (1):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03448510/Prot_000.pdf